CLINICAL TRIAL: NCT04374201
Title: Fourteen-year Evaluation of Posterior Zirconia-based Three-unit Fixed Dental Prostheses. A Prospective Clinical Study of All Ceramic Prosthesis
Brief Title: 14y Prospective Study on Posterior Zirconia-based 3-unit FDPs
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Fernando Zarone, Professor, Federico II University
Other Study IDs: 3Y-TZP Federico II
Record Dates: First submitted 2020-04-24; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Prosthesis Survival
Keywords: zirconia; all ceramic prosthesis; prosthodontics; fixed dental prosthesis; prosthetic dentistry; prospective clinical study
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2 zirconia FDPs: 11 patients received 2 zirconia fixed dental prostheses
  Interventions: Other: 2 zirconia FDPs
- 1 zirconia FDP: 26 patients received 1 zirconia FDP
  Interventions: Other: 1 zirconia FDP

INTERVENTIONS:
Other: 2 zirconia FDPs — The United States Public Health Service criteria were used in order to examine technical and esthetic outcomes. Success and survival rates of the zirconia FDPs were calculated. The biological examination was performed analyzing both abutments and contralateral teeth.
  Groups: 2 zirconia FDPs
Other: 1 zirconia FDP — The United States Public Health Service criteria were used in order to examine technical and esthetic outcomes. Success and survival rates of the zirconia FDPs were calculated. The biological examination was performed analyzing both abutments and contralateral teeth.
  Groups: 1 zirconia FDP

SUMMARY:
The main objective of the present prospective study is to evaluate the effectiveness of posterior zirconia FDPs after 14 years of function.

DETAILED DESCRIPTION:
thirty-seven patients needing to replace either premolars or molars were involved and 48 3-unit zirconia-based FDPs were fabricated. Patients included in the present clinical study met specific inclusion criteria and clinical procedures were standardized.

Frameworks with a 9 mm2 cross section of the connectors and 0.6 mm minimum thickness of the retainers were made by means of Computer Aided Design/Computer Assisted Manufacturing. A resin cement was used to lute the restorations. The patients were recalled after 6 and 12 months and then yearly up to a total follow-up of 14 years. The United States Public Health Service criteria were used in order to examine technical and esthetic outcomes. Success and survival rates

ELIGIBILITY:
Inclusion Criteria:

* good general health;
* ASA I or ASA II according to the American Society of Anesthesiologists;
* good periodontal health;
* Angle class I occlusal relationship;
* minimum of 20 teeth;
* good oral hygiene;
* no evident signs of occlusal parafunctions and/or temporo-mandibular disorders.

Moreover, the abutment teeth had to fulfill the following inclusion criteria:

* periodontal health (absence of tooth mobility, absence of furcation involvement);
* proper positioning in the dental arch (tooth axes adequate for a FDP);
* sufficient occlusal-cervical height of the clinical crown (≥4 mm) for the retention of a FDP;
* vital or endodontically treated to a clinically sound state;
* opposing natural teeth or fixed prostheses.

Exclusion Criteria:- subjects preferring implant-supported prostheses;

* high caries activity;
* occlusal-gingival height of the abutment teeth <4 mm;
* reduced interocclusal distance or supraerupted opposing teeth;
* unfavorable crown-to-root ratio;
* severe wear facets, clenching, bruxism;
* presence of removable partial dentures;
* pregnancy or lactation.

Ages: 21 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the present prospective clinical study, 37 patients (16 males, 21 females) needing at least 1 posterior FDP in the maxillary and/or the mandibular arches were recruited. The mean age of patients was 45.3 ± 11.6 years, with a minimum age of 21 and a maximum of 68 years. All patients were recruited at the Department of Prosthodontics of the University "Federico II" of Naples (Italy) from November 2004 to April 2005 (baseline) and provided a written informed consent
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2004-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival and success rate of zirconia FDPs | 14 years
  The 14-year cumulative survival rate of the zirconia FDPs was calculated by means of Kaplan-Meier analysis.

SECONDARY OUTCOMES:
Technical and aesthetic outcomes | 14 years
  The United States Public Health Service criteria were used in order to examine technical and esthetic outcomes.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT04374201/Prot_SAP_000.pdf